CLINICAL TRIAL: NCT05722067
Title: Improved the Low Fertilization Rates and Increased the High-quality Embryogenesis by Treatment with Calcium Ionophore GM508 CultActive Optimized Medium in Vitro Fertilization (IVF) Patients
Brief Title: Improvement of Fertilization Rate and Embryo Quality by Treating Calcium Ionophore in IVF Patients: a Sibling Oocyte Control Study
Acronym: GM508 in IVF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202200969A3
Record Dates: First submitted 2022-11-20; First posted 2023-02-10 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: IVF; Infertility; Artificial Oocyte Activation
Keywords: artificial oocyte activation; calcium ionophore; ivf; poor responder
MeSH Terms: conditions — Infertility; Long Qt Syndrome 3 | interventions — Calcium Ionophores

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oocytes treated with calcium ionophore (Experimental): Oocytes treated with a ready-to-use ionophore compound (GM508 CultActive, Gynemed) within 15 min after ICSI (or 18 min in IVF). After 15 min of incubation in GM508 CultActive and a thorough washing process, the oocytes subjected to AOA will transfer to the same time-lapse culture dish with the controlled sibling group.
  Interventions: Other: calcium ionophore
- oocytes undergo routine IVF/ICSI protocol (No Intervention): Untreated control oocytes will immediately place into the time-lapse imaging system, and the culture protocol was routine.

INTERVENTIONS:
Other: calcium ionophore — The intervention group will be treated with a ready-to-use ionophore medium (GM508 CultActive, Gynemed) within 15 min after ICSI (or 18 min in IVF) based on the situation of sperm. After 15 min of incubation in GM508 CultActive and a thorough washing process, the oocytes will be cultured in the same protocol as the control group.
  Other Names: GM508 CultActive
  Arms: oocytes treated with calcium ionophore

SUMMARY:
GM508 CultActive is a bicarbonate buffered reagent and ready-to-use designed to investigate oocytes of patients with failed fertilization after previous Intracytoplasmatic Sperm Injection cycles. The investigators hypothesize that GM508 CultActive will improve the fertilization rate and embryo development of such IVF patients (a history of poor fertilization, a history of poor embryo quality, and over 40 years old expected challenging to conceive).

ELIGIBILITY:
Inclusion Criteria:

* Low fertilization rate in previous IVF cycle (<30%), or
* Poor embryo developmental problems in previous IVF cycle, or
* Diminished ovarian reserve (AMH<1.2 or AFC<5) and/or more than 40 y/o.

Exclusion Criteria:

* Without or just one oocyte picked up

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
fertilization rate | Day 1
  The normal fertilization rate will defined as the number of zygotes with 2PN and 2PB per the total number of mature oocytes

SECONDARY OUTCOMES:
blastocyst formation rate | Day 5
  NO. of blastocysts per 2PN zygotes
top-quality blastocyst formation rate | Day 5
  No. of 3AA, 4AA, 5AA or 6AA blastocysts / 2PN zygotes
pregnancy outcome | 1 year
  pregnancy rates, abortion rate, live birth rates,congenital anomaly rate

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No